CLINICAL TRIAL: NCT01218919
Title: A CLINICAL EVALUATION OF A RECHARGEABLE DEEP BRAIN STIMULATION SYSTEM AS AN ADJUNCTIVE TREATMENT FOR REDUCING SOME OF THE SYMPTOMS OF ADVANCED, LEVODOPA-RESPONSIVE PARKINSON'S DISEASE THAT ARE NOT ADEQUATELY CONTROLLED WITH MEDICATION
Brief Title: Post Market (Brio™ System) Deep Brain Stimulation (DBS) PD Study
Status: Withdrawn | Type: Observational
Why Stopped: Business reasons
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-10-017-ID-DB
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Brio DBS System: Eligible subjects in this study will be screened to confirm that they meet the strict guidelines for advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication followed by bilateral surgery to implant the Brio™ deep brain stimulation system

SUMMARY:
The objective of this study is to evaluate the effectiveness of a rechargeable Deep Brain Stimulation as an adjunctive treatment for reducing some of the symptoms of advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication.

This is the first observational study for the use of the BRIO™ rechargeable constant current device, using a lead with an active electrode tip for deep brain stimulation in Parkinson subjects. The current study was designed to conform to normal medical practices, taking into consideration the current day economic constraints, while assessing the best set of circumstances for the successful sustained reduction of some of the symptoms of advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational, non-randomized, multi-centered study for a total of 10 years in duration. It is a 10 year study from system implantation and activation with a yearly database lock and report, with the subjects being used as their own control. The primary outcome assessment will occur at three months. Following completion of the primary outcome assessment, patients will have an annual visit up to 10 years post implant.

Comparison of measures within the same person from pre-treatment to post-treatment will be performed.

During the implantation procedure, each subject will undergo a trial of stimulation in the operating room among other potential assessments to determine proper lead placement. The device may be internalized after a successful intra-operative trial or at a later date according to investigator site practice. The date that all components are implanted and programmed will be classified as "Day 0". After system activation the subject will return to clinic for post-operative evaluations at 1 month (+/-14 days), 3 months (+/-14 days), 6 months (+/-14 days) and 12 months (+/-30 days). Thereafter, a long term data collection program will be followed for 10 years post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an informed consent.
2. Subject has been diagnosed, by a neurologist, with idiopathic Parkinson's disease.
3. Subject is a candidate for surgery.
4. Subject is 18 to 80 years of age.
5. Subject has a history of improvement of Parkinson's symptoms as a direct result of administering L-dopa to the subject with at least a 25% improvement in UPDRS motor score or subject has been diagnosed with tremor-dominant Parkinson's disease.
6. Subject should be stable on anti-Parkinson's disease medication for at least one month prior to study enrollment

Exclusion Criteria:

1. Subject has any major illness or medical condition that in the opinion of the physician would interfere with participation in the study.
2. Subject has non-treated clinically significant depression or any other significant psychiatric co-morbidities.
3. Subject has any condition requiring repeated MRI scans;
4. Subject is on anticoagulant medications and is unable to interrupt for time of procedure.
5. Subject has dementia that interferes with their ability to co-operate or comply with study requirements or comprehend the Informed Consent as determined by the investigator.
6. Subject abuses drugs or alcohol.
7. Subject has a history of seizure (Neurosurgeon must approve)
8. Subject has confirmation of diagnosis of a terminal illness associated with survival <12 months.
9. Female that is lactating or of childbearing potential with positive urine pregnancy test or not using adequate birth control.
10. Subject has participated in a drug, device or biological trial within the preceding 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication
  Eligible subjects in this study will be screened to confirm that they meet the strict guidelines for advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
UPDRS motor scores | 3 months after device implantation
  Comparison of Parkinson's symptoms as demonstrated by the UPDRS motor scores in the medication 'Off' state at Baseline compared to the medication 'Off' with stimulation "On" 3 months after device implantation

SECONDARY OUTCOMES:
PDQ-8 | 3, 6 and 12 months compared to baseline
  Quality of Life measurements through 3, 6 and 12 months as measured by the PDQ-8 compared to baseline
modified Schwab and England | 3, 6 and 12 months compared to baseline
  Activities of Daily Living measurement through 3, 6 and 12 months as determined from the modified Schwab and England, compared to baseline
Levodopa dose | baseline and 3, 6 and 12 month after device implantation
  Comparison of Levodopa dose taken by the subject at baseline and 3, 6 and 12 month after device implantation
Satisfaction of therapy | 3, 6 and 12 months
  Rate of subject and caregivers therapy satisfaction through 3, 6 and 12 months
IPG Recharging information | 3 and 12 months
  Evaluation of the subjects/caregivers IPG Recharging information